CLINICAL TRIAL: NCT06201481
Title: Clinical Success of Anterior and Posterior Full Coverage Restorations in a Group of Children Treated Under General Anesthesia: An Incidence Study
Brief Title: Clinical Success of Anterior and Posterior Crowns in a Group of Children Treated Under General Anesthesia
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Salma Sayed Ali Ebrahim, Principal Investigator, Cairo University
Other Study IDs: Success in Dental GA
Record Dates: First submitted 2023-12-16; First posted 2024-01-11 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Prosthesis Failure, Dental
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: anterior and posterior full coverage crowns — Teeth preparation,crown fitting and cementation

SUMMARY:
* This incidence study aims to evaluate the clinical success of anterior and posterior full-coverage restorations among a group of Egyptian children treated under general anesthesia.
* The main question it aims to answer:

In A Group of Children, What Is the Clinical Success of Anterior and Posterior Full Coverage Restorations Performed Under General Anesthesia?

DETAILED DESCRIPTION:
This study consisted of clinical examinations of the participants treated under general anesthesia to evaluate the clinical success of anterior and posterior crowns that will be performed on the day of the dental treatment, then after 15 days, 3, 6, and 12 months recall examinations.

- The level of parental satisfaction will be evaluated through a questionnaire that will be completed after 15 days, 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 2 and 5 years old.
* Children classified as American Society of Anesthesiologists class I; Healthy (no acute or chronic disease, normal BMI percentile for age)
* All Children received pulp therapy techniques for vital teeth.

Exclusion Criteria:

* Children with mental or neurological disorders.
* Children with developmental disorders and syndromes.
* Children whose parents have no mobile phone access.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Egyptian Children Aged 2-5 years.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Clinical Success of Stainless-Steel Crowns | Immediately after the intervention then after 15 days then after 3 months then after 6 months and after 12 months
  Clinical evaluation criteria:
  * crown marginal adaptation
  * crown marginal extension crown proximal contact
  * duration of crown presence
Clinical Success of Anterior Esthetic Crowns | Immediately after the intervention then after 15 days then after 3 months then after 6 months and after 12 months
  Clinical evaluation criteria:
  * crown retention
  * crown chipping
  * opposing wear

SECONDARY OUTCOMES:
Pain score | Immediately after the intervention then after 15 days then after 3 months then after 6 months and after 12 months
  Pain will be evaluated by scores using a five-point scale.
  * None (If the parents give a score 1)
  * Mild (If the parents give a score 2)
  * Moderate (If the parents give a score 3)
  * Sever (If the parents give a score 4 or 5)

OTHER OUTCOMES:
Level of Parental Satisfaction | After 15 days of the Intervention then after 3 months then after 6 months and after 12 months
  A questionnaire will measure the level of parental satisfaction.
  - Questions will be answered by YES or NO .
  The questions :
  * Received enough information before treatment?
  * Knew where and how to access help after treatment?
  * Regarded this treatment to be positive?
  * Overall experience is satisfactory?
  * Would consider general anesthesia for treatment again?

REFERENCES:
- [Background] Schuler IM, Hiller M, Roloff T, Kuhnisch J, Heinrich-Weltzien R. Clinical success of stainless steel crowns placed under general anaesthesia in primary molars: an observational follow up study. J Dent. 2014 Nov;42(11):1396-403. doi: 10.1016/j.jdent.2014.06.009. Epub 2014 Jun 30. PMID 24994618
- [Result] Jiang H, Shen L, Qin D, He S, Wang J. Effects of dental general anaesthesia treatment on early childhood caries: a prospective cohort study in China. BMJ Open. 2019 Sep 9;9(9):e028931. doi: 10.1136/bmjopen-2019-028931. PMID 31501107
- [Result] Sharaf AA, Farsi NM. A clinical and radiographic evaluation of stainless steel crowns for primary molars. J Dent. 2004 Jan;32(1):27-33. doi: 10.1016/s0300-5712(03)00136-2. PMID 14659715
- [Result] MacLean JK, Champagne CE, Waggoner WF, Ditmyer MM, Casamassimo P. Clinical outcomes for primary anterior teeth treated with preveneered stainless steel crowns. Pediatr Dent. 2007 Sep-Oct;29(5):377-81. PMID 18027771
- [Result] Chao Z, Gui Jin H, Cong Y. The effect of general anesthesia for ambulatory dental treatment on children in Chongqing, Southwest China. Paediatr Anaesth. 2017 Jan;27(1):98-105. doi: 10.1111/pan.12983. Epub 2016 Oct 25. PMID 27779347